CLINICAL TRIAL: NCT00202501
Title: Usefulness of Nasal CPAP Treatment in Patients With a First Ever Stroke and Sleep Apnea Syndrome
Brief Title: Usefulness of Nasal Continuous Positive Airway Pressure (CPAP) Treatment in Patients With a First Ever Stroke and Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: PII Sueño SEPAR
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI030184
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Sleep Apnea; Stroke; Cardiovascular Disease
MeSH Terms: conditions — Sleep Apnea Syndromes; Stroke; Cardiovascular Diseases | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Nasal CPAP (Continuous Positive Airway Pressure)

SUMMARY:
MAIN AIMS: to analyze the efficacy of nasal CPAP treatment in patients with ischemic first-ever stroke and Sleep Apnea Syndrome (SAS) in terms of: early neurological outcome, functional recovery, quality of life influence, stroke recurrence and survival.

SECONDARY AIMS: to evaluate the feasibility of the treatment in this type of patients at short and long time.

DESIGN: clinical randomized case-control study.

PATIENTS: younger than 75 years with a First-Ever stroke with at least one of the following criteria: snoring, observed apnea, Hypertension or Ischemic Cardiopathy.

MEASUREMENTS: protocol to define subtype stroke and parenchymatous and vascular location; sleep questionnaire (including Epworth Sleepiness Scale); Respiratory Polysomnography (RPSG). If RPSG shows an AHI > 20, with predominant obstructive events, patients will be randomized in a CONTROL GROUP (conventional treatment) and a TREATMENT GROUP (with Nasal CPAP). Follow up for both groups at 1, 3, 12 and 24 months will include: early neurological outcome, body mass index (BMI), blood pressure (BP), functional recovery (Barthel Index/Canadian Scale), quality of life (SF36), recurrences, vital status. Nasal CPAP titration will be performed by means of an automatic system (Autoset Portable ST). Compliance will be recorded. If a negative RPSG is obtained (AHI < 10) (NO SAS GROUP) or with AHI < 20 (mild SAS) the usual treatment and the same follow up protocol will be established.

STATISTICS: the sample size is initially calculated in 10 patients for each group, considering this is part of a multicenter study including 8 centers. If no differences are found, depending on the statistical power the investigators will consider including more patients. The different groups will be compared for the analyzed variables with the corresponding tests.

ELIGIBILITY:
Inclusion Criteria:

* First ever stroke
* Any Sleep Apnea symptom
* Hypertension

Exclusion Criteria:

* Aphasia
* Cognitive impairment
* Hypersomnolence

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2006-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Neurologic recovering
Quality of life
Recurrences

SECONDARY OUTCOMES:
To assess feasibility of Nasal CPAP treatment in patients with stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Parra, MD, Principal Investigator — Hospital Universitari Sagrat Cor
Locations (1):
- Hospital Universitari Sagrat Cor, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Reynor A, McArdle N, Shenoy B, Dhaliwal SS, Rea SC, Walsh J, Eastwood PR, Maddison K, Hillman DR, Ling I, Keenan BT, Maislin G, Magalang U, Pack AI, Mazzotti DR, Lee CH, Singh B. Continuous positive airway pressure and adverse cardiovascular events in obstructive sleep apnea: are participants of randomized trials representative of sleep clinic patients? Sleep. 2022 Apr 11;45(4):zsab264. doi: 10.1093/sleep/zsab264. PMID 34739082
- [Derived] Parra O, Sanchez-Armengol A, Bonnin M, Arboix A, Campos-Rodriguez F, Perez-Ronchel J, Duran-Cantolla J, de la Torre G, Gonzalez Marcos JR, de la Pena M, Carmen Jimenez M, Masa F, Casado I, Luz Alonso M, Macarron JL. Early treatment of obstructive apnoea and stroke outcome: a randomised controlled trial. Eur Respir J. 2011 May;37(5):1128-36. doi: 10.1183/09031936.00034410. Epub 2010 Sep 16. PMID 20847081